CLINICAL TRIAL: NCT00022243
Title: A Phase II, Open Label Study Of T138067-Sodium In A Second-Line Setting In Non-Small-Cell Lung Cancer Patients With Locally Advanced Or Metastatic Disease Who Have Failed First-Line Therapy With a Taxane
Brief Title: T138067 in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer That Has Not Responded to Previous Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tularik (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068798; TULA-T2002; VU-000511
Record Dates: First submitted 2001-08-10; First posted 2004-02-04 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Drug: batabulin sodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of T138067 in treating patients who have locally advanced or metastatic non-small cell lung cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective tumor response rate in patients with locally advanced or metastatic non-small cell lung cancer who have failed first-line therapy with a taxane when treated with T138067 sodium. II. Determine the qualitative and quantitative toxic effects of this drug in these patients. III. Determine the number of patients who progress when treated with this drug. IV. Determine the duration of response, time to disease progression, and median survival of patients treated with this drug. V. Correlate the toxic effects of this drug with peak plasma levels in this patient population.

OUTLINE: This is a multicenter study. Patients receive T138067 sodium IV over 3 hours on days 1, 8, and 15. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months after study completion.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed non-small cell lung cancer (NSCLC) Locally advanced or metastatic disease Received a prior first-line taxane (as a single agent or component of a combination regimen) as the only chemotherapy for locally advanced or metastatic disease Any amount of prior adjuvant chemotherapy allowed Bidimensionally measurable disease outside the field of prior radiotherapy Amenable to radiologic imaging techniques No clinically apparent CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST and ALT no greater than 3 times ULN Albumin greater than 2.5 g/dL No history of Gilbert's syndrome Renal: Creatinine no greater than 1.5 times ULN Other: No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No other severe disease, infection, or comorbidity that would preclude study participation No known defect of glutathione metabolism Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy or therapeutic biologic response modifiers No concurrent routine or prophylactic filgrastim (G-CSF) or sargramostim No concurrent epoetin alfa Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered No other concurrent cytotoxic chemotherapy Endocrine therapy: No concurrent hormonal therapy for NSCLC Radiotherapy: See Disease Characteristics At least 2 weeks since prior limited-field radiotherapy not involving the hematopoietic bone marrow and recovered At least 4 weeks since prior radiotherapy to no more than 25% of the hematopoietic bone marrow and recovered No prior wide-field radiotherapy to the pelvis No concurrent radiotherapy (including palliative radiotherapy) Surgery: At least 4 weeks since prior major surgery Other: At least 4 weeks since prior investigational agents No concurrent anticonvulsants unless required for study drug-related toxicity No concurrent high-dose acetaminophen (i.e., at least 4 g/day) No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Sean McCarthy, Study Chair — Tularik
Locations (2):
- United States (2):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Jahan TM, Sandler A, Burris H, et al.: A phase II study of T138067-sodium in prior taxane-treated patients (pts) with locally advanced or metastatic non-small cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1282, 2002.